CLINICAL TRIAL: NCT00976768
Title: A Phase II Study of Biweekly Oxaliplatin and 5-Fluorouracil/Leucovorin Combination Chemotherapy (FOLFIRI) in Patients With Advanced Gastric Cancer (AGC) With Failure of Prior Chemotherapy Including Taxane, Fluoropyrimidine and Cisplatinum
Brief Title: Biweekly FOLFIRI in Advanced Gastric Cancer (AGC) With Failure of Prior Taxane, Fluoropyrimidine, and Cisplatin
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yoon-Koo Kang, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC0402
Record Dates: First submitted 2009-09-11; First posted 2009-09-14 (Estimated); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Advanced Gastric Cancer
Keywords: Advanced gastric cancer; FOLFIRI
MeSH Terms: interventions — Oxaliplatin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFIRI arm (Experimental): Patients receiving FOLFIRI
  Interventions: Drug: oxaliplatin, 5-fluorouracil

INTERVENTIONS:
Drug: oxaliplatin, 5-fluorouracil — Oxaliplatin 85 mg/㎡ IV, day 1 over 2 hours 5-FU 400 mg/㎡ IV bolus day 1 followed by 5-fluorouracil(FU) 2,400 mg/㎡ and leucovorin (LV) 100 mg/㎡ IV continuous over 46 hours (every 2 weeks)

SUMMARY:
The purpose of this study is:

* To observe the feasibility of biweekly oxaliplatin and infusional 5-fluorouracil (FU)/Leucovorin (LV) in patients with advanced gastric adenocarcinoma who have prior exposure to taxane, fluoropyrimidine, and cisplatin
* To determine the activity of this combination regimen.
* To evaluate the treatment-related toxicities.

DETAILED DESCRIPTION:
There is presently no chemotherapy regimen considered to be the standard of care for patients with advanced gastric cancer. However, more and more patients will receive fluoropyrimidine, platinum, and taxane combination or sequential chemotherapy. Unfortunately, about half of the patients receiving chemotherapy are unresponsive and treatment results of salvage chemotherapy are unsatisfactory. For these patients, there are currently no established palliative chemotherapy options, and there is urgent need for novel, active, and less toxic regimens for patients with advanced gastric cancer failing front-line chemotherapy.

On these bases, we will investigate the activity of biweekly oxaliplatin and 5-FU/LV in patients with advanced gastric cancer who failed prior taxane, fluoropyrimidine and cisplatin chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically proven non-resectable adenocarcinoma of stomach
* Measurable disease based on Response Criteria in Solid Tumors (RECIST)
* Prior chemotherapy with taxane, fluoropyrimidine, and cisplatinum in combination or sequentially, there is no time limit for the last chemotherapy
* Age 18 to 70 years old
* Estimated life expectancy of more than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 2 or lower
* Adequate bone marrow function (white blood cell counts >4,000/µL, absolute neutrophil count [ANC]>1,500/µL, hemoglobin >9.0 g/dL, and platelets>100,000/µL),
* Adequate kidney function (creatinine<1.5 mg/dL)
* Adequate liver function (bilirubin<1.5 mg/dL , transaminases levels<3 times the upper normal limit [5 times for patients with liver metastasis], and serum albumin of >2.5 mg/dL)

Exclusion Criteria:

* Other tumor type than adenocarcinoma
* Presence or history of central nervous system metastasis
* Obvious or impending bowel obstruction (including obvious peritoneal carcinomatosis)
* Evidence of active gastrointestinal bleeding
* Other serious illness or medical conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | 4 months

SECONDARY OUTCOMES:
Overall survival | 1 year
Toxicity profile (according to National Cancer Institute Common Terminology Criteria for Adverse Event [NCI CTC AE] version 3.0) | Each cycle of chemotherapy
Response rate | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan medical center, Seoul, South Korea